CLINICAL TRIAL: NCT02291978
Title: A Feasibility Study to Evaluate the Safety and Initial Effectiveness of MR Guided High Intensity Focused Ultrasound (MRgHIFU) in the Treatment of Facetogenic Lumbar Back Pain
Brief Title: MR Guided High Intensity Focused Ultrasound for Lumbar Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients met eligibility.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Pejman Ghanouni, Assistant Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29163
Record Dates: First submitted 2014-11-05; First posted 2014-11-17 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Lumbar Facet Joint Pain
Keywords: back pain; facet joint; spine
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ExAblate 2100 Treatment (Experimental): The ExAblate 2100 system will be used in the MRgHIFU treatment of lower back pain arising from facet joint arthritis.
  Interventions: Device: ExAblate 2100

INTERVENTIONS:
Device: ExAblate 2100 — The InSightec ExAblate 2100 MRgHIFU system is a non-invasive thermal ablation device fully integrated with an MR imaging system and used for the ablation of soft tissue and bone.

SUMMARY:
The primary purpose of this protocol is to assess the ExAblate 2100 MR guided high intensity focused ultrasound device as an intervention for treatment of facetogenic lower back pain.

DETAILED DESCRIPTION:
This is a single group, single arm, open/nonblinded, non-randomized study. The primary outcomes are safety and preliminary efficacy. The InSightec ExAblate 2100 MRgHIFU system is a non-invasive thermal ablation device fully integrated with an MR imaging system and used for the ablation of soft tissue and bone.The study will reach primary completion 12 months from the time the study opens to accrual.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women > 21 years of age and who are skeletally mature
2. Body mass index ≤ 30 kg/m2
3. Patients who are able to understand and willing to sign a written informed consent document and able to attend all study visits
4. Patients with at least 6 months of chronic lower back pain (LBP) localized to the midline or axial low back, with symptoms attributed to the facet joints on physical examination that have persisted despite conservative therapy. Conservative therapy is defined as systemic pain medications and anti-inflammatory medications, as well as physical therapy, such as massage, heating, hydrotherapy, and strengthening exercises.
5. Patients with Numerical Rating Scale worst lumbar back pain score of at least 4 out of 10 over the 24 hours preceding the time of rating.
6. Patients must have chronic LBP attributed to facet joints as demonstrated by MRI consistent with at least grade 2 facet joint arthritis, with corresponding abnormal activity at the facet joint on 18F-sodium fluoride PET-CT.
7. Patients must have an analgesic response to either prior local anesthetic injection to the facet joint or to radiofrequency ablation of the facet joint, with relapse of pain.
8. The targeted facet joint must be deeper than 10 mm from the skin

Exclusion Criteria:

1. Patients with severe lumbar lordosis
2. Patients with contraindication for MR imaging such as implanted metallic devices that are not MRI-safe, size limitations, claustrophobia. etc
3. Patients with known intolerance or allergy to MR contrast agent (gadolinium chelates) including advanced kidney disease (GFR <30 mL/min/1.73 m2) or on dialysis
4. Pregnant and nursing patients will be excluded from the study because of a contraindication to administering MRI contrast agents to these patients
5. Patients with known intolerance or allergy to medications used for sedation (midazolam), analgesia (fentanyl), and local and regional anesthesia (lidocaine, bupivacaine, and ropivacaine)
6. Patients with evidence of lumbosacral radiculopathy on MRI or physical exam findings, including radicular leg pain, or any neurologic deficit at or below the segmental level of the highest facet to be treated, including subjects with impaired sphincter control
7. Patients with pain at another location that

   1. cannot be distinguished from lumbar back pain
   2. does not rate at least 2 points less in worst pain score compared to lumbar back pain
   3. requires the use of analgesics
8. Patients with gross spinal instability on imaging
9. Patients who have lumbar spinal stabilization hardware in place
10. Target is:

    * NOT visible by non-contrast MRI, OR
    * NOT accessible to ExAblate device
11. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (can be up to 5 hrs of total table time)
12. Patients with acute medical condition (e.g. pneumonia, sepsis) that is expected to hinder them from completing this study
13. Patients with unstable cardiac status including:

    1. Unstable angina pectoris on medication
    2. Patients with documented myocardial infarction within six months of protocol entry
    3. Congestive heart failure requiring medication (other than diuretic)
    4. Patients on anti-arrhythmic drugs
14. Patients with severe hypertension (diastolic BP > 100 on medication)
15. Patients with severe hematologic, neurologic, or other uncontrolled disease (e.g. platelets < 50,000/microL, INR > 1.5)
16. Patients who are taking anti-thrombotic medication
17. Severe cerebrovascular disease (multiple CVAs or CVA within 6 months)
18. Patients with inflammatory arthritides.
19. Patients unable to communicate with the investigator and staff
20. Patients seeking compensation for disability or work injury.
21. Patients who are part of another trial testing other Investigational Agents

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Device Related Complications as a Measure of Safety | 24 months
  Safety will be determined by evaluating for the incidence and severity of any device related complication from the treatment day visit through 24 months after treatment.

SECONDARY OUTCOMES:
Pain Relief on the Visual Analog Scale | 24 months
  Effectiveness will be determined by the level of pain relief, as measured by the NRS, and decrease in analgesic/opiate use.
Quality of Life Improvement | 24 months
  Effectiveness will be determined by improved quality of life, as measured by the Oswestry Disability Index.

CONTACTS AND LOCATIONS:
Overall Officials: Pejman Ghanouni, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States